CLINICAL TRIAL: NCT01052116
Title: The Study of Soy Isoflavones in Asthma
Acronym: SOYA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: American Lung Association Asthma Clinical Research Centers (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Robert A. Wise, M.D., Director of Data Coordinating Center, American Lung Association Asthma Clinical Research Centers
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ALAACRC-10; R01HL087987-01A2 (Other: NIH/NHLBI); R01 HL0088367-01A2 (Other: NIH/NHLBI)
Record Dates: First submitted 2009-12-04; First posted 2010-01-20 (Estimated); Results first posted 2016-01-14 (Estimated); Last update posted 2016-01-14 (Estimated); Status verified 2015-12

CONDITIONS: Asthma
Keywords: Asthma; Soy; Supplement; ACRC; SOYA
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Soy Isoflavone (Active Comparator): Oral isoflavone supplement (100 mg/day)
  Interventions: Drug: Soy isoflavone supplement
- Placebo (Placebo Comparator): Matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Soy isoflavone supplement — Oral soy isoflavone supplement (100 mg/day)
  Other Names: Soy supplement
  Arms: Soy Isoflavone
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The trial is designed to study the effects of soy supplements on asthma control.

DETAILED DESCRIPTION:
Asthma is a common disease that has a major impact on morbidity and health care costs. Although the prevalence and severity of asthma have increased over the last several decades, the specific causes remain unknown. One possible mechanism is a change in diet. Yet, epidemiological and interventional studies designed to identify a key nutrient or antioxidant vitamin that may be responsible for the increase in disease severity have produced inconsistent results. A recent pilot study showed a soy isoflavone supplement reduces exhaled nitric oxide (FeNO) and ex vivo LTC4 synthesis in patients with inadequately controlled asthma. This clinical trial is designed to test the novel hypothesis that dietary supplementation with soy isoflavones is an effective treatment in patients with poorly controlled asthma. The study will include 380 patients with low dietary soy intake, 12 years of age or older, who are taking either inhaled corticosteroids or leukotriene modifiers and have inadequately controlled asthma. Participants will be randomly assigned to treatment with either a soy isoflavone supplement (containing genistein, daidzein and glycitein; 100 mg daily of the glycoside forms) or placebo for six months. The results of this trial will increase understanding of the role of diet in asthma; could identify a novel, safe and relatively inexpensive treatment for patients with asthma; and potentially will have a substantial impact on public health in the United States.

ELIGIBILITY:
Inclusion Criteria:

* Age 12 or older
* Physician diagnosed asthma

  * FEV1 equal or greater than 50% predicted pre-bronchodilator
  * At least 12% increase in FEV1 15-3 minutes after inhaling 2-4 puffs of albuterol or positive methacholine challenge (20% fall in FEV1 at less than 8 mg/mL). Either of these can be available from the previous 2 years
  * Currently prescribed daily controller asthma medication
* Poor asthma control (at least one of the following)

  * A score of 1.5 or greater on the Juniper Asthma Control Questionnaire
  * Use of beta-agonist for asthma symptoms two or more times per week
  * Nocturnal awakening with asthma symptoms more than once per week
  * Two or more episodes of asthma symptoms in the past 12 months with each requiring at least one of the following: emergency department visit, unscheduled physician visit, prednisone course, hospitalization
* Smoking status

  * Non-smoker for 6 months or longer
  * Less than 10 pack-years smoking history

Exclusion Criteria:

* Pulmonary function

  * FEV1 less than 50% predicted pre-bronchodilator
* Other major chronic illnesses

  * Conditions which in the judgment of the study physician would interfere with participation in the study, e.g., non-skin cancer, endocrine disease, coronary artery disease, severe hypertension, immunodeficiency states
  * History of thyroid disease, breast cancer, ovarian, or endometrial cancer
  * History of physician diagnosis of chronic bronchitis, emphysema, or COPD
* Medication use

  * Current consumption of soy isoflavone supplements
  * Oral corticosteroid use within the past 6 weeks
  * Use of tamoxifen
* Use of an investigational treatment in the previous 30 days
* "Drug" allergy

  * Known adverse reaction to genistein, other phytoestrogens, or soy products
* Females of childbearing potential

  * Pregnant or lactating. Participants must agree to use effective contraception during the trial.
* Non-adherence

  * Inability or unwillingness to provide consent or, in the case of children, inability or unwillingness of the child to provide assent
  * Inability to swallow study medication
  * Inability to perform baseline measurements
  * Completion of less than 10 of the last 14 days diary entries during screening period
  * Inability to be contacted by telephone
  * Intention to move out of the area within 6 months
* Other

  * Recent asthma exacerbation (within 6 weeks)
  * Recent upper respiratory infection (within 2 weeks)
  * Body weight less than 77 pounds (35 kg)
  * Intake of soy or soy-enriched foods 1 or more times a week
  * Change in diet over the past month or expected change in diet during the study

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 386 (Actual)
Dates: Start 2010-03; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lewis J Smith, MD, Principal Investigator — Northwestern University
Locations (18):
- United States (18):
  - University of Arizona, Tucson, Arizona
  - University of California, San Diego, San Diego, California
  - National Jewish Health, Denver, Colorado
  - Nemours Children's Clinic, Jacksonville, Florida
  - University of Miami School of Medicine, Miami, Florida
  - University of South Florida College of Medicine, Tampa, Florida
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - Louisiana State University Health Sciences Center, New Orleans, Louisiana
  - University of Missouri, Kansas City School of Medicine, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - North Shore - Long Island Jewish Health System, New Hyde Park, New York
  - New York University School of Medicine, New York, New York
  - New York Medical College, Valhalla, New York
  - Duke University Medical Center, Durham, North Carolina
  - Davis Heart and Lung Research Institute, Columbus, Ohio
  - Baylor College of Medicine, Houston, Texas
  - Vermont Lung Center at the University of Vermont, Burlington, Vermont

REFERENCES:
- [Result] Smith LJ, Kalhan R, Wise RA, Sugar EA, Lima JJ, Irvin CG, Dozor AJ, Holbrook JT; American Lung Association Asthma Clinical Research Centers. Effect of a soy isoflavone supplement on lung function and clinical outcomes in patients with poorly controlled asthma: a randomized clinical trial. JAMA. 2015 May 26;313(20):2033-43. doi: 10.1001/jama.2015.5024. PMID 26010632
- [Derived] Kaminsky DA, He J, Henderson R, Dixon AE, Irvin CG, Mastronarde J, Smith LJ, Sugar EA, Wise RA, Holbrook JT. Bronchodilator response does not associate with asthma control or symptom burden among patients with poorly controlled asthma. Respir Med. 2023 Nov;218:107375. doi: 10.1016/j.rmed.2023.107375. Epub 2023 Aug 1. PMID 37536444
- See also: ALA-ACRC Webpage — http://www.cctrials.org/alaacrc

RESULTS

PARTICIPANT FLOW:
Groups:
- Soy Isoflavone: Oral soy isoflavone supplement
  Tablet twice a day (100 mg/day)
Period: Overall Study
Arm/Group | Placebo | Soy Isoflavone
Started | 193 | 193
Completed | 179 (Completed: defined as having an FEV1 measurement at 24 weeks) | 166 (Completed: defined as having an FEV1 measurement at 24 weeks)
Not Completed | 14 | 27
Not completed — Lost to Follow-up | 11 | 17
Not completed — Withdrawal by Subject | 3 | 6
Not completed — Spirometry not performed | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Matching placebo
  Tablet twice a day
- Total: Total of all reporting groups
Arm/Group | Placebo | Soy Isoflavone | Total
Number analyzed (Participants) | 193 | 193 | 386
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 38 [17 to 49] | 34 [20 to 49] | 36 [18 to 49]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 125 | 129 | 254
  Male | 68 | 64 | 132
FEV1 [Median (Inter-Quartile Range); unit: Liters] | 2.44 [1.96 to 2.93] | 2.40 [2.01 to 2.91] | 2.43 [1.99 to 2.91]

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline to 24 Weeks for FEV1
Time Frame: 24 weeks
Measure: Mean (95% Confidence Interval); unit: Liters
Groups:
- Soy Isoflavone: Oral soy isoflavone supplement
  tablet twice daily (100 mg/day)
- Placebo: Matching placebo
  Tablet twice daily
Arm/Group | Soy Isoflavone | Placebo
Number analyzed (Participants) | 193 | 193
Liters | -0.001 [-0.07 to 0.07] | 0.03 [-0.01 to 0.08]

ADVERSE EVENTS:
Time Frame: trial conducted for 2 years each participant followed for 24 weeks
Arm/Group | Placebo | Soy Isoflavone
Serious Adverse Events (participants affected / at risk) | 12/193 | 12/193
Other Adverse Events (participants affected / at risk) | 130/186 | 132/186
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=193) | Soy Isoflavone (N=193)
Pulmonary including asthma exacerbation (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 3 (3)
Cardiovascular, circulatory, and lymphatic (Cardiac disorders) | 0 (0) | 1 (1)
Renal/urinary (Renal and urinary disorders) | 1 (1) | 0 (0)
Gastrointestinal (Gastrointestinal disorders) | 0 (0) | 2 (4)
Neuropsychiatric (Nervous system disorders) | 0 (0) | 4 (4)
Reproductive (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Integumentary (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Placebo (N=186) | Soy Isoflavone (N=186)
Rash (Skin and subcutaneous tissue disorders) | 40/160 | 39/167
Itching (Skin and subcutaneous tissue disorders) | 45/139 | 47/147
Difficulty breathing (Respiratory, thoracic and mediastinal disorders) | 47/77 | 48/81
Difficulty swallowing (Gastrointestinal disorders) | 38/179 | 31/171
Hypotension (Blood and lymphatic system disorders) | 10/182 | 14/180
Breast tenderness (Musculoskeletal and connective tissue disorders) | 24/180 | 21/175
Change in menstrual symptoms (Reproductive system and breast disorders) | 33/62 | 43/71

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No